CLINICAL TRIAL: NCT05743569
Title: Virtual Patient-specific 3D Specimen Maps for Adjuvant Head & Neck Radiotherapy Planning
Brief Title: 3D Specimen Maps for RT Planning
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Topf, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 222115
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Radiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this study is to measure the impact of patient-specific 3D specimen maps on adjuvant radiation treatment volumes and doses to critical organs. All patients will receive standard-of-care post-operative radiotherapy not impacted by the experimental 3D specimen maps. The secondary objective is to demonstrate the feasibility of incorporating 3D specimen mapping tools into post-operative communication, and to determine if utilization of the 3D specimen map improves post-operative communication between surgeons, pathologists, and radiation oncologists.

DETAILED DESCRIPTION:
It is estimated that 65,000 new cases of head and neck squamous cell carcinoma (HNSCC) were diagnosed in the United States in 2020. The incidence of HNSCC is projected to increase 30% worldwide by 2030. Surgical resection is the preferred treatment for oral cavity cancer and frequently plays a role in the management of oropharyngeal and laryngeal cancer. Approximately 70-80% of patients who undergo primary resection for oropharyngeal HNSCC will receive post-operative radiotherapy. Post-operative radiotherapy is generally indicated for HNSCC with features associated with high risk of locoregional recurrence, such as stage pT3 or pT4 primary tumors, close or positive margins, multiple involved lymph nodes, extranodal extension, or the presence of multiple additional high risk features such as lymphovascular invasion, perineural invasion, deep depth of invasion, or high grade.

The delineation of post-operative target volumes for localization and radiation planning can be difficult for the treating radiation oncologist due to post-operative anatomy changes from surgical manipulation of tissues, loss of normal tissue planes, and post-operative fluid collections. Post-operative radiotherapy treatment plans and volumes are usually delineated by the radiation oncologist based on review of a combination of data points including operative reports, pre-operative and post-operative diagnostic images, pathology reports, identification of surgical clips, and discussions with the treating head and neck surgeon and/or pathologists. Generally, the post-operative Clinical Target Volume for the primary tumor (CTVp) should include the primary tumor operative bed with a suitable margin to account for microscopic spread and is generally treated to 60Gy. For tumors with a positive margin, some radiation oncologists may choose to boost the area of positive margin up to 66Gy. The CTV boost (CTVb) can be difficult to visualize, and accurate understanding of the location of the positive margin can influence how small or large the boost volume is and thus dose to adjacent normal tissues, or organs at risk (OARs).

Optical 3D scanning technology has been a standard procedure quality control in industrial manufacturing for years. Due to its speed, accuracy, and relative ease of use, 3D scanning has steadily proven its utility in medicine over the past decade. The investigators have developed a protocol for optical 3D scanning of the specimen to improve communication between the OR and pathology lab (Figure 2). The resected specimen is scanned using a structured light 3D scanner. Graphics software is then used to virtually ink and annotate 3D specimen models, indicating and clearly defining the specific anatomic locations of the frozen section margins (Figure 3). In the present study, the investigators aim to use the patient-specific 3D specimen maps to improve communication between surgeons and radiation oncologists for adjuvant radiation therapy treatment planning and determine the impact of these 3D specimen maps on CTVs and OARs.

3D innovations are numerous and have become a well-established avenue of research in otolaryngology and a variety of other fields over the past decade. Optical innovations increasingly represent a new diagnostic modality that has demonstrated potential for intraoperative guidance.The team of investigators has previously published a study on the use of 3D scanning technology and virtual graphics software to bridge the gap between the operating room and pathology lab. The investigators determined this relatively simple, non-invasive technique to be a valuable communication tool for surgeons and pathologists responsible for the care of patients with head and neck cancer. However, the utilization of this technology in post-operative discussions and treatment planning with radiation oncologists has yet to be evaluated. The overarching goal of this research is to improve communication and mutual comprehension between the surgeon, pathologist, and radiation oncologist using commercially available, readily implementable 3D scanning technology and virtual graphics software thus to improve delineation of post-operative radiation therapy target volumes for patients with head and neck cancer.

The primary objective of this study is to measure the impact of patient-specific 3D specimen maps on adjuvant radiation treatment volumes and doses to critical organs. All patients will receive standard-of-care post-operative radiotherapy not impacted by the experimental 3D specimen maps. The secondary objective is to demonstrate the feasibility of incorporating 3D specimen mapping tools into post-operative communication, and to determine if utilization of the 3D specimen map improves post-operative communication between surgeons, pathologists, and radiation oncologists.

Aim #1 - Measure the impact of patient-specific 3D specimen maps on adjuvant radiation treatment fields The investigators hypothesize that the use of virtual 3D specimen mapping in radiation treatment planning will impact clinical target volumes (CTVs) to the primary tumor bed (CTVp) and/or boost (CTVb) and doses to adjacent organs at risk because of improved understanding of gross and microscopic tumor involvement.

The investigators will compare volume measurements between CTVs of two radiation treatment plans: one using standard of care planning techniques and the other with the addition of virtual 3D specimen mapping. The investigators will also compare radiotherapy doses to determine any changes to adjacent organs at risk between the two radiation treatment plans. All patients will be treated with the standard of care radiation plan that does not incorporate the 3D specimen tool.

Aim #2 - Investigate the subjective benefit of 3D specimen mapping on postoperative communication with the radiation oncologist.

The investigators hypothesize that 3D scanning and specimen mapping will benefit key stakeholders (surgeons, pathologists, radiation oncologists). Surveys will be administered at baseline and at the end of the study to assess the perceived effect of the 3D specimen tool on post-operative communication of pathology relevant to radiation field design (ie, location of positive or close margins, orientation of gross tumor in specimen, volume of resected specimen, etc).

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. Biopsy-confirmed mucosal head and neck cancer. All histologic malignancies will be included.
3. Patients who have completed primary tumor surgical resection in the following anatomic subsites:

   1. oral cavity (oral tongue, floor of mouth, hard palate, buccal mucosa, retromolar trigone, maxillary and mandibular alveolus, lip)
   2. oropharynx (soft palate, base of tongue, palatine tonsils)
   3. hypopharynx (piriform sinus, post-cricoid, posterior pharyngeal wall)
   4. larynx (supraglottic, glottic, subglottic);
4. Patients who have consented to 3D specimen mapping on protocol IRB # 221597 and for whom 3D specimen maps are therefore available.
5. Patients are indicated to receive curative-intent post-operative radiotherapy and intend to receive radiotherapy at Vanderbilt University Medical Center or Vanderbilt Ingram Cancer Center sites in Nashville, Franklin, or Lebanon

Exclusion Criteria:

1. Under the age of 18
2. Cutaneous malignancies
3. Characteristics that make the process of informed consent questionable
4. Pregnant women
5. Patients with contraindications to radiotherapy

Min Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to recruit adult patients with biopsy-confirmed mucosal head and neck cancer who have completed primary tumor surgical resection of their cancer.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Measure the impact of patient-specific 3D specimen maps on adjuvant radiation treatment fields | 1 year
  The investigators hypothesize that the use of virtual 3D specimen mapping in radiation treatment planning will impact clinical target volumes (CTVs) to the primary tumor bed (CTVp) and/or boost (CTVb) and doses to adjacent organs at risk because of improved understanding of gross and microscopic tumor involvement.
  The investigators will compare volume measurements between CTVs of two radiation treatment plans: one using standard of care planning techniques and the other with the addition of virtual 3D specimen mapping. The investigators will also compare radiotherapy doses to determine any changes to adjacent organs at risk between the two radiation treatment plans. All patients will be treated with the standard of care radiation plan that does not incorporate the 3D specimen tool.

SECONDARY OUTCOMES:
Investigate the subjective benefit of 3D specimen mapping on postoperative communication with the radiation oncologist. | 1 year
  The investigators hypothesize that 3D scanning and specimen mapping will benefit key stakeholders (surgeons, pathologists, radiation oncologists). Surveys will be administered at baseline and at the end of the study to assess the perceived effect of the 3D specimen tool on post-operative communication of pathology relevant to radiation field design (ie, location of positive or close margins, orientation of gross tumor in specimen, volume of resected specimen, etc).

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States